CLINICAL TRIAL: NCT02726659
Title: Adjunctive Use of Celecoxib in the Treatment of Bipolar Postpartum Depression: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Adjunctive Use of Celecoxib in the Treatment of Bipolar Postpartum Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty recruiting participants because principal investigator noticed that the participants in the population were responding well to low doses of mood stabilizers and therefor would not be recruited into the study.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 107775
Record Dates: First submitted 2016-03-15; First posted 2016-04-04 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2018-11

CONDITIONS: Bipolar Disorder; Postpartum Depression
MeSH Terms: conditions — Bipolar Disorder; Depression, Postpartum | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celecoxib (Experimental): Adjunct celecoxib in 6 week treatment
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Adjunct placebo in 6 week treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Adjunct celecoxib
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Placebo — Adjunct placebo
  Arms: Placebo

SUMMARY:
The investigators will conduct a 6-week, randomized, double-blind, placebo-controlled trial of celecoxib as an add-on treatment to the mood stabilizer among women with bipolar I or II postpartum depression. Women who are taking a mood stabilizer for treatment of bipolar disorder in the postpartum treatment will receive either a placebo or celecoxib add-on treatment. Patients will be monitored regularly to assess psychiatric symptoms and side effects. The investigators aim to evaluate the potential antidepressant effect of celecoxib in bipolar postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-45 who are within 3 months of delivering a healthy, term (37 to 40 weeks) singleton
* diagnosis of bipolar postpartum depression - depressed with peripartum onset
* have a 17-item Hamilton Rating Scale for Depression score of >18
* have failed to respond to an adequate trial of the mood stabilizer
* are currently not on any psychotropic drug except a mood stabilizer (lithium, lamotrigine or quetiapine)
* are able to communicate (written and oral) in English and capable of giving consent

Exclusion Criteria:

* current major depressive episode of more than 6 months duration
* a current comorbid psychiatric disorder
* history of alcohol or substance abuse within the 12 months before screening
* concurrent psychotherapy
* high risk for suicide (actively suicidal or a score of = 3 on item #3 on HAM-D)
* current hepatic, renal, or cardiac disease, chronic pain, coagulation disorders, esophageal or gastro duodenal ulceration within the previous 30 days
* known immediate-type hypersensitivity to COX-2 inhibitors, sulfonamides, ibuprofen, or diclofenac
* breastfeeding mothers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | 6 weeks
  To assess the effectiveness of the addition of celecoxib in the treatment of bipolar postpartum depression by the change in mean scores on the HAM-D between baseline and the 6 weeks endpoint. Response will be a > 50% reduction in HAM-D score and remission will be a < 7 HAM-D score from baseline to week 6.

SECONDARY OUTCOMES:
Montgomery Asberg Depression Scale | 6 weeks
  To assess the effectiveness of the addition of celecoxib in the treatment of bipolar postpartum depression as measured by the change in the mean scores on the Montgomery Asberg Depression Rating Scale between baseline and the study termination endpoint.
Udvalg for Kliniske Undersogelser Scale | 6 weeks
  To assess the tolerability of celecoxib in women with bipolar postpartum depression as assessed by the Udvalg for Kliniske Undersogelser Scale.
Edinburgh Postnatal Depression Scale (EPDS) | 6 weeks
  To assess the effectiveness of the addition of celecoxib in the treatment of bipolar postpartum depression as measured by the mean change in scores on the EPDS between baseline and the study termination endpoint.
Clinical Global Impression Scale (CGI) | 6 weeks
  To assess the effectiveness of the addition of celecoxib in the treatment of bipolar postpartum depression as measured by the change in scores on the CGI between baseline and the study termination endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Verinder Sharma, MB BS, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Parkwood Institute, Mental Health Care Buildling, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
A data sharing agreement will be in place between Lawson Health Research Institute and The National Institute for Mental Health Research.